CLINICAL TRIAL: NCT00632879
Title: The Study of Metabolic Syndrome in Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Shao-Yu Yang/Attending Physician, Far Eastern Memorial Hospital and National Taiwan University Hospital
Other Study IDs: 96011
Record Dates: First submitted 2008-03-03; First posted 2008-03-11 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-07

CONDITIONS: Hemodialysis; Metabolic Syndrome X; Insulin Resistance
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are collected for analysis

SUMMARY:
Metabolic syndrome (MS), comprised of central obesity, glucose intolerance, hyperinsulinemia, low HDL-cholesterol (HDL-C), high triglyceride (TG) and hypertension, results in markedly increased risk for cardiovascular disease in the general population. The National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) report recommended the use of five variables for the diagnosis of the MS including waist circumference (WC), serum TG concentration, serum HDL-C concentration, blood pressure and fasting glucose concentration. A waist circumference of 80 cm in women and 90 cm in men would better identify those with the MS in Asian populations. However, the studies of modified asian criteria of metabolic syndrome in hemodialysis (HD) patients are scarce.

We will perform prevalence investigation, cross-sectional study, and prospective investigation for metabolic syndrome in our HD patients (around 360 at present). We will enroll all the patients who receive maintenance HD more than three months in our HD center. The patients who are hospitalizing, suffered from active malignancy, active infections, recent cardiovascular events and surgery will be excluded in the beginning of study. Biochemistry and anthropometric parameters including HDL-C, TG, insulin resistance index, high sensitivity C-reactive protein and WC will be collected and analyzed. We will also prospectively establish the mortality and hospitalization indices of these patients, to study the prognosis of HD patient with or without metabolic syndrome.

This study will be helpful to understand whether the application of a modified criteria of metabolic syndrome in HD patients is capable to predict cardiovascular events, hospitalization and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* We will enroll all the patients who receive maintenance HD more than three months in our HD center.

Exclusion Criteria:

* The patients who are hospitalizing, suffered from active malignancy, active infections, recent cardiovascular events and surgery will be excluded in the beginning of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive maintenance hemodialysis in our HD center
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-03; Study Completion 2008-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Yu Yang, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, PanChiao, Taipei, Taiwan